CLINICAL TRIAL: NCT03398967
Title: Phase I/II Study to Evaluate Treatment of Relapsed or Refractory Leukemia and Lymphoma With Universal CRISPR-Cas9 Gene-Editing CAR-T Cells Targeting CD19 and CD20 or CD22
Brief Title: A Feasibility and Safety Study of Universal Dual Specificity CD19 and CD20 or CD22 CAR-T Cell Immunotherapy for Relapsed or Refractory Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Molecular & Immunological Department, Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-026
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: B Cell Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Universal Dual Specificity CD19 and CD20 or CD22 CAR-T Cells — 1. Biological: Universal Dual Specificity CD19 and CD20 or CD22 CAR-T Cells
  2. Day 0: 10% of total dose Day 1: 30% of total dose if patient is stable (no significant toxicity) from prior dose. D2: 60% of total dose if patient is stable (no significant toxicity) from prior dose
  3. Other: Laboratory Biomarker Analysis

SUMMARY:
CD19-directed CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory B-cell malignancies; however, a subset of patients relapse due to the loss of CD19 in tumor cells. Dual Specificity CD19 and CD20 or CD22 CAR-T cells can recognize and kill the CD19 negative malignant cells through recognition of CD20 or CD22. This is a phase 1/2 study designed to determine the safety of the allogenic gene-edited dual specificity CD19 and CD20 or CD22 CAR-T cells and the feasibility of making enough to treat patients with relapsed or refractory hematological malignancies.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVES:

   1. To evaluate the feasibility and safety of universal dual specificity CD19 and CD20 or CD22 CAR-T cells in patients with relapsed or refractory leukemia and lymphoma.
   2. To evaluate the duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells. Real Time polymerase chain receptor (RT-PCR) and Flow cytometry(FCM) analysis of PB,BM and lymph node will be used to detect and quantify survival of universal dual specificity CD19 and CD20 or CD22 CAR-T cells over time.
2. SECONDARY OBJECTIVES:

   1. For patients with detectable disease, measure anti-tumor response due to universal dual specificity CD19 and CD20 or CD22 CAR-T cell infusions.
   2. Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable universal dual specificity CD19 and CD20 or CD22 CAR-T cells (loss of engraftment).

The CAR-T cells will be administered by i.v. injection over 20-30 minutes as a using a "split dose" approach to dosing: 10% on day 0, 30% on day 1 and 60% on day 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant
2. 12 Years to 70 Years (Child, Adult, Senior)
3. Patient with relapsed or refractory B-cell leukemia or lymphoma
4. Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Adequate organ function

Exclusion Criteria:

1. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
2. Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis
3. Richter's syndrome
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
5. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
6. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
7. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
8. Patient has an investigational medicinal product within the last 30 days prior to screening
9. Previous treatment with investigational gene or cell therapy medicine products
10. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
11. Pregnant or nursing women

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety and Tolerability | 24 weeks
MTD of universal dual specificity CD19 and CD20 or CD22 CAR-T cells | 4 weeks
  The highest dose of universal dual specificity CD19 and CD20 or CD22 CAR-T cells that is estimated to result in defined Dose Limiting Toxicity (DLT) with the exception of allowable 'expected' AEs associated with the intravenous infusion of universal dual s
Copies numbers of CAR in peripheral blood(PB), bone marrow(BM)and lymph nodes | 24 weeks

SECONDARY OUTCOMES:
Six-month Objective response rate of complete remission and partial remission | 24 weeks
Six-month Overall survival | 24 weeks
Six-month Progression free survival | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China